CLINICAL TRIAL: NCT00013312
Title: Effects of Acute SCI on Colonic Motility & Tone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B1862R
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury, gastrointestinal motility, gastrointestinal transit
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Procedure: Determine colonic tone

SUMMARY:
This study will compare individuals with acute SCI to control patients in order to: 1. Determine if there are changes in colonic tone and sensation after SCI by comparing the fasting responses to the postprandial responses; 2. Determine if there are changes in colonic phasic motility after SCI by comparing the fasting responses to the postprandial responses; 3. Determine if colonic motor and sensory function after SCI change over time by repeating these studies six month later in SCI and control patients.

ELIGIBILITY:
Acute SCI with impaired colonic tone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 1999-04; Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D. Asst. Director — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Nancy Rocheleau, Program Analyst — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, Hines, Hines, Illinois, United States